CLINICAL TRIAL: NCT04793841
Title: Population Burden of Sexually Transmitted Infections and Implication for Intervention in Hong Kong
Brief Title: Population Burden of STI and Implication for Intervention in Hong Kong
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ngai Sze WONG, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: CID-CUHK-E
Record Dates: First submitted 2021-02-01; First posted 2021-03-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: STI
Keywords: chlamydia trachomatis; Neisseria gonorrhoeae; human papillomavirus; men who have sex with men; general population
MeSH Terms: conditions — Sexually Transmitted Diseases; Homosexuality | interventions — Laboratories

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, penile swab, cervical swab, rectal swab, pharyngeal swab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population: sexually experienced adults (aged 18 or above) of the randomly selected household
  Interventions: Other: self-sampling kits for STI testing in laboratory
- men who have sex with men: men who have sex with men aged 18 or above and normally living in Hong Kong
  Interventions: Other: self-sampling kits for STI testing in laboratory

INTERVENTIONS:
Other: self-sampling kits for STI testing in laboratory — participants in both groups will receive self-sampling kits and deliver the collected samples to laboratory for testing

SUMMARY:
This is a 5-year cross-disciplinary sexually transmitted infection (STI) project involving a) territory-wide and community-based studies (survey and specimen collection); b) simulation of STI transmission dynamics and comparison of STI intervention strategies through mathematical modelling and cost-effectiveness analysis. The aim of this project is to assess the burden and the transmission dynamics of STIs in the general population and men who have sex with men (MSM) in Hong Kong. Around 1300 sexually experienced adults and 900 MSM would be recruited, 100 participants would be invited for individual in-depth interviews. Main outcome measures include STI history and service preference, effectiveness as measured by the proportion of new STI infections (chlamydia, gonorrhoea and human papillomavirus infections) averted above base-case scenario, and incremental cost-effectiveness ratio.

DETAILED DESCRIPTION:
After completion of baseline questionnaire, the participants are invitied for STI self-sampling. If agree, a package of self-sampling kits, instructions, and packaging materials for return post would be delivered to their selected collection points. The second round of self-sampling would be offered at least one year from the first round of self-sampled specimens collected.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* ever having sex
* normally living in Hong Kong
* can communicate in English or Chinese

Exclusion Criteria:

* failed to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: sexually experienced adults
Sampling Method: Probability Sample
Enrollment: 1977 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
self-reported STI diagnosis in questionnaire | up to 2 years
  number of STI diagnosis
effectiveness of STI intervention strategies | 10 years
  incremental cost-effectiveness ratio

SECONDARY OUTCOMES:
STI symptom reported in questionnaire | 12 months
  types of symptom presentations
willingness to pay for STI testing reported in questionnaire | 12 months
  willingness to pay (HKD)
prevalence of STI estimated through laboratory testing | 12 months
  prevalence of chlamydia trachomatis, Neisseria gonorrhoeae and human papillomavirus infections from self-collected samples

CONTACTS AND LOCATIONS:
Overall Officials: Ngai Sze Wong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong, China, Hong Kong

IPD SHARING:
Plan to Share IPD: No